CLINICAL TRIAL: NCT02251028
Title: Value-based Cognitive Behavioural Therapy for the Prevention of Chronic Whiplash Associated Disorders: A Randomized Controlled Trial
Brief Title: Value-based Cognitive Behavioral Therapy for Prevention of Chronic Whiplash-associated Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Tonny Elmose Andersen, phd., MSc., Ph.D, University of Southern Denmark
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: S-20130103
Record Dates: First submitted 2014-09-19; First posted 2014-09-26 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Musculoskeletal Disorders; Whiplash
Keywords: whiplash, prevention, pain, cognitive-behavioural therapy
MeSH Terms: conditions — Musculoskeletal Diseases; Whiplash Injuries; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): Group A receives value-based cognitive behavior therapy after randomization.
  Interventions: Behavioral: Value-based cognitive-behavioral therapy
- Group B (Active Comparator): Group B receives value-based cognitive behavior therapy after 3 months.
  Interventions: Behavioral: Value-based cognitive-behavioral therapy

INTERVENTIONS:
Behavioral: Value-based cognitive-behavioral therapy — The intervention is a manualized program specifically tailored for prevention of disability and psychological distress after whiplash injuries. The intervention is delivered by two trained clinical psychologists og consists of 10 weekly one-hour individual sessions.

SUMMARY:
The purpose of this study is to determine whether a specifically tailored value-based cognitive behavioural therapy program (V-CBT) is able to prevent the development of persistent disability, pain, and psychological distress if delivered within the first three months after a whiplash injury.

DETAILED DESCRIPTION:
The primary objective of the present study is to test whether a specifically tailored value-based cognitive-behavioural therapy program (V-CBT) is able to prevent the development of persistent disability, pain, and psychological distress if delivered within the first three months after a whiplash injury. Methods. The current study is a two-armed randomized controlled study with a crossover design. Group A is scheduled for V-CBT within one week of randomization and group B with a delayed onset 3 months after randomization.

ELIGIBILITY:
* 18 and 65-years-old
* WAD level I-II.
* 3-months post-injury
* Disability in at least one important life domain (≥ 5 on the pain disability index) and moderate levels of pain (average pain intensity ≥ 4 on the NRS scale).
* Meet at least one of the psychological risk criteria:
* Elevated levels of pain catastrophizing, fear-avoidance-beliefs, symptoms of anxiety and/or depression, and posttraumatic stress symptoms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Disability as measured by Pain Disability Index | Change scores at 12- and 24-weeks after randomization
  The PDI measures how pain interferes with daily life activities within 7 different domains. The 7 domains are rated from 0 (no disability) to 10 (worst disability). The scale shows good reliability and validity.

SECONDARY OUTCOMES:
Pain by NDI | Change scores at 12- and 24-weeks after randomization
  Neck pain intensity and disability is measured with the Neck Disability Index (NDI; Vernon & Mior, 1991). The NDI measures within 10 domains pain and how neck pain affects the ability to handle daily life activities such as personal care, lifting, reading, work, driving, sleeping, recreational activities, pain intensity, concentration, and headache. The total score range from 0 (no disability) to 100 (total disability).
Pain by NRS | Change scores at 12- and 24-weeks after randomization
  Pain is also measured on four numerical pain rating scales (NRS) ranging from 0 (no pain) to 10 (worst possible pain). Patients mark their answers on each scale corresponding to their pain now, highest level of pain, lowest level of pain, and finally average pain over the past week (NRS: Turk & Melzack, 2001).
Fear of re-injury by TSK | Change scores at 12- and 24-weeks after randomization
  Fear of re-injury due to movement is measured with Tampa Scale for Kinesiophobia (TSK; Kori, Miller, & Todd, 1990). TSK is a 17-item scale assessing fear of movement on a 4-point likert scale ranging from 17 to 68 with higher scores indicating higher levels of kinesiophobia. The scale is commonly used in various chronic pain samples and has good construct and predictive validity (Roelofs, Goubert, Peters, Vlayen, & Crombes, 2004). The clinical cut-off score is set to ≥ 37.
Pain-related catastrophizing by PCS | Change scores at 12- and 24-weeks after randomization
  Catastrophic thinking related to pain is measured with the Pain Catastrophizing Scale (PCS; Sullivan, Bishop, Pivik, 1995). The PCS-instructions ask participants to reflect on past painful experiences and to indicate the degree to which they experienced each of 13 thoughts or feelings when experiencing pain on a five-point Likert scale with (0 = not at all, 4 = all the time).
Anxiety and depression by HADS | Change scores at 12- and 24-weeks after randomization
  To assess the level of anxiety and depressive symptoms, the Hospital Anxiety and Depression Scale is used (HADS; Zigmond & Snaith, 1983). The scale consists of 14 items, 7 relating to anxiety (HADS-A) and 7 to depression (HADS-D) with responses ranging from 0 (no symptoms) to 3 (maximum impairment). A cut-off score of ≥ 8 on each subscale is used in order to include all possible cases of depression and anxiety as suggested by (Zigmond & Snaith, 1983).
PTSD-symptomatology | Change scores at 12- and 24-weeks after randomization
  PTSD-symptomatology is measured with the PTSD-8 (Hansen, Andersen, Armour, Elklit, Palic, & Mackrill, 2010). The scale is a brief version of The Harvard Trauma Questionnaire part IV (HTQ-IV; Molicca, Caspi-Yavin, Bollini, & Truong, 1992) and consists of 8 items on a four-point Likert scale (1 = not at all, 4 = very often). The items relate to the three core clusters in PTSD in DSM-IV: avoidance (2 items), intrusion (4 items), and hyperarousal (2 items). The scale has proven good psychometric properties in various trauma samples including whiplash injured (Hansen et al., 2010).

CONTACTS AND LOCATIONS:
Overall Officials: Tonny Elmose Andersen, MSc,Ph.D., Study Director — Department of Psychology; Ask Elklit, professor, Study Director — Department of Psychology
Locations (1):
- University of Southern Denmark, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersen TE, Ravn SL, Roessler KK. Value-based cognitive-behavioural therapy for the prevention of chronic whiplash associated disorders: protocol of a randomized controlled trial. BMC Musculoskelet Disord. 2015 Sep 1;16:232. doi: 10.1186/s12891-015-0687-y. PMID 26323830